## **Informed Consent to Participate in Research**

## BMT CTN 1401 v4.0

Phase II Multicenter Trial of Single Autologous Hematopoietic Cell Transplant Followed by Lenalidomide Maintenance for Multiple Myeloma with or without Vaccination with Dendritic Cell /Myeloma Fusions

| Your Name: | |
|---|---|
| Study Title: | Phase II Multicenter Trial of Single Autologous Hematopoietic Cell<br>Transplant Followed by Lenalidomide Maintenance for Multiple Myeloma<br>with or without Vaccination with Dendritic Cell /Myeloma Fusions |
| Protocol: | BMT CTN 1401 v4.0 |
| Principal<br>Investigator: | Insert local PI information |
| Sponsor: | The National Institutes of Health (NIH) is sponsoring this study by providing financial support for the coordination of this study through the Blood and Marrow Transplant Clinical Trials Network (BMT CTN). |

## 1. Introduction

We invite you to join this clinical trial, also known as a research study. You are being asked to join because:

- You're  $\geq$ 18 and <71 years old
- You have multiple myeloma (MM)
- Your doctor thinks an **autologous transplant** is a possible treatment option for you.

The standard of care for patients with MM is an autologous transplant and **maintenance treatment**. Maintenance treatment is chemotherapy after transplant. There's no cure for MM, so patients get maintenance treatment to slow the return of MM after a transplant.

We're doing this study to learn if maintenance treatment works better alone or with a vaccine made from your own blood cells.

This study will take at least 3 years and will include 203 participants. Your participation will last for a maximum of 4 years from when you are enrolled.

This consent form will tell you about the purpose of the study, the possible risks and benefits, other options available to you, and your rights as a participant in the study.

Everyone who takes part in research at [insert facility name] should know that:

- Being in any research study is voluntary.
- You may or may not benefit from being in the study. Knowledge we gain from this study may benefit others.
- If you join the study, you can quit the study at any time.
- If you decide to quit the study, it will not affect your care at [insert name of facility or institution].
- Please ask the study staff questions about anything that you do not understand, or if you would like to have more information.
- You can ask questions now or any time during the study.

• Please take the time you need to talk about the study with your doctor, study staff, and your family and friends. It is your decision to be in the study. If you decide to join, please sign and date the end of the Consent Form.

You and your doctor will discuss other treatment choices if you do not want to participate in this study.

## 2. Study Background

The National Institutes of Health (NIH), through the Blood and Marrow Transplant Clinical Trials Network (BMT CTN), are providing staff support and money for this research study. The BMT CTN and the NIH will make decisions about how to manage the study.

For this study, you will receive an **autologous transplant** (transplant). An autologous transplant uses blood-forming cells that are collected from your blood stream. After they are collected and frozen, you will get a high dose of chemotherapy. Chemotherapy before a transplant is called the "conditioning regimen".

The goal of chemotherapy is to kill as many cancer cells in your body as possible. It also destroys most of the normal cells in your bone marrow. To restore your marrow, your frozen blood-forming cells are thawed and transplanted back into your blood stream. The cells find their way into the bone marrow where they start making healthy blood-forming cells.

The standard of care for patients with MM is an autologous transplant and **maintenance treatment**. Maintenance treatment is chemotherapy after transplant. There's no cure for MM, so patients get maintenance treatment to slow the return of MM after a transplant.

Some patients may receive a vaccine, and/or GM-CSF (also known as Leukine) with their maintenance therapy. GM-CSF helps your body make new white blood cells after transplant.

The vaccine is made from dendritic cells and MM tumor cells in a laboratory. We will collect a sample of your cells through your central line (or catheter). This process is called leukapheresis. If the vaccine is made successfully, it will be frozen and stored to give to you later.

We're doing this study to learn if maintenance treatment works better alone, or with a vaccine made from your own blood cells.

## 3. Study Purpose

We are inviting you to take part in this study because you have multiple myeloma (MM) and an autologous transplant is a treatment option for you. We are doing this study to learn more about ways to prevent or slow the return of MM after transplant.

We will use 3 treatments to see which one works best to prevent or slow the return of MM. See **Table 1** for information on each treatment group.

**Table 1. Study Treatment Groups** 

| Treatment Group A (maintenance treatment with GM-CSF <u>and</u> vaccines) | Treatment Group B (maintenance treatment with GM-CSF) | Treatment Group C (only maintenance treatment) |
|---|---|---|
| <ul> <li>Melphalan (chemotherapy drug)</li> <li>Autologous transplant</li> <li>Lenalidomide (maintenance treatment)</li> <li>GM-CSF</li> <li>Vaccine</li> </ul> | <ul> <li>Melphalan (chemotherapy drug)</li> <li>Autologous transplant</li> <li>Lenalidomide (maintenance treatment)</li> <li>GM-CSF</li> </ul> | <ul> <li>Melphalan (chemotherapy drug)</li> <li>Autologous transplant</li> <li>Lenalidomide (maintenance treatment)</li> </ul> |

This study will help doctors make the best choice about treatment after transplant for patients with MM. See section **5: Study Tests and Treatments** for information on how your treatment group will be determined and for information about the drugs listed in **Table 1**.

# 4. Rights to Ask Questions and/or Withdraw

You have the right to ask questions about the study at any time. If you have questions about your rights as a participant or you want to leave the study, please contact:

[insert contact info]

Being in this study is voluntary. You can choose not to be in this study or leave this study at any time. If you choose not to take part or leave this study, it will not affect your regular medical care in any way.

Your study doctor and study staff will be available to answer any questions that you may have about taking part in or leaving this study.

# 5. Study Treatment and Tests

We will check your health <u>before</u> you start treatment, <u>during</u> your treatment, and for <u>3 years after</u> you begin your maintenance treatment.

#### **Before You Start Your Treatment**

You will need to have several check-ups and tests to see if you can be in the study. These check-ups and tests are part of your regular cancer care and would be done even if you were not part of this study. These tests include:

- Medical history and physical exam
- Blood tests for cell counts
- Liver and kidney function tests
- Tests to measure your disease
- Bone marrow tests
- Skeletal survey
- A pregnancy test (if you are a woman able to have children)

#### **During Your Treatment**

#### **Tumor Cell Collection**

After you join the study, we will collect about 30mL (approximately 2 tablespoons) of bone marrow and 50mL (approximately 3 tablespoons) of blood. The bone marrow and blood samples will be frozen until it is determined if you will receive the vaccine as part of your treatment. This tumor cell collection is not part of your standard of care treatment

If you are assigned to Treatment Group A after your transplant, your bone marrow will be thawed and used to make your vaccine. If you are assigned to Treatment Group B or C, your

bone marrow sample will not be used in this study. Your doctor may talk to you about other uses for your stored bone marrow samples not related to this study.

We will also talk with you about giving extra blood and marrow samples for future research (see section 17: Blood and Marrow Samples for Future Research). The extra blood and marrow samples are also completely optional.

## <u>Initial Treatment for Multiple Myeloma (MM)</u>

The first step (initial) is standard chemotherapy treatment (chemo). Chemo lowers the number of MM cells in your body. Different chemotherapy drugs can be used to treat MM. Your doctor will decide which drug or combination of drugs is best for you.

You will be asked to sign a separate consent form that will explain the side effects of whichever drug your doctor chooses. This step may last several months.

#### **Blood-Forming Cell Collection**

Next, we'll collect blood-forming cells from your blood stream. This is known as apheresis. These cells will be frozen and stored until your transplant day.

## Conditioning Regimen Before Transplant

The third step is the conditioning regimen, or the <u>chemotherapy</u>, you will get before your transplant. The conditioning regimen helps the blood-forming cells start to grow and make new cells in your bone marrow (engraft). The regimen includes a chemo drug called **melphalan**, given by intravenous infusion (IV) in your arm.

Your doctor will decide when you are ready to get melphalan. You will start this treatment step no more than 12 months after you start on this study. Melphalan works better for some patients than it does for others. If the drug does not work well for you, you may not be able to have a transplant. Your doctor will talk to you about other treatment options.

## <u>Infusion of Blood Forming Cells (Transplant)</u>

On your transplant day (Day 0), your cells will be given to you through your catheter. The cells will travel to your bone marrow where they will start to make healthy, new blood cells (engraft).

#### Your Treatment Group

Approximately 2 months after transplant, we will check to see if you're healthy enough to start maintenance treatment. If you are found healthy enough, we will randomize you to 1 of the 3 treatment groups. "Randomize" means that you will be put in one or another group by chance, just like flipping a coin. We will use a computer program to assign you by chance to Treatment

Group A, B, or C. You won't be able to choose your group. Once you are assigned to a group, you can't change to another group. The study doctor can't change your group either.

Half of the patients on this study (about 66), will be assigned to Treatment Group A. One-fourth of the patients (about 33) will be assigned to Treatment Group B; and one-fourth of patients (about 33) will be assigned to Treatment Group C. See the section below, **Your Maintenance**Treatment After Transplant, for a description of the treatments.

Once all these tests are done, you will be randomized to Treatment Group A, B or C. See **Table 2** for a schedule of these tests.

If you're not healthy enough after transplant, you won't be randomized. If this happens, your Follow up on this study is complete

#### Your Maintenance Treatment After Transplant

You will start maintenance treatment about 3 months after your transplant.

#### > Treatment Group A: Lenalidomide, Vaccine, and GM-CSF injections

If you are assigned to Treatment Group A, you will get: lenalidomide, vaccines, and GM-CSF injections.

We will collect extra blood samples to make the vaccine. We will insert a catheter into a large vein in your neck or chest. The catheter will collect some blood cells and the rest are returned to your body. This process is called leukapheresis. We will use the blood cells and the marrow that was collected and frozen to create your vaccine. The vaccine will be made in a laboratory and frozen until you're ready for maintenance treatment.

You will take lenalidomide as a pill every day for 2 years or until your disease returns. You will receive enough pills for 1 cycle (28 days in each cycle) at a time. It's important to take the pill at the same time every day. Be sure to talk with your doctor to figure out a good time to take the pill every day.

You will also receive 3 doses of the vaccine. This will be given to you on the first day of your 2<sup>nd</sup>, 3<sup>rd</sup>, and 4<sup>th</sup> cycle of lenalidomide. The vaccine is the part of the treatment we are testing in this study. This is also called the research treatment.

With each vaccine, you will also get an injection of GM-CSF in your upper thigh. GM-CSF helps to boost the effect of the vaccine. You will receive the GM-CSF injection on the day you get the vaccine and every day for 3 days after the vaccine. This will either be given to you in the clinic or you will be taught to give the injections to yourself at home.

See **Table 2** for a timeline of the drugs for Treatment Group A.

**Table 2: Treatment Group A** 

| | | | Timeline for Maintenance Treatment Drugs | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group A<br>drugs: | Amount: | Cycle:<br>(28 days<br>in each<br>cycle) | 1 | 2 | 3 | 4 | 6 | 9 | 12 | 15 | 18 | 21 | 24 |
| Lenalidomide | 1 dose eve<br>2 ye | | X | X | X | X | X | X | X | X | X | X | X |
| Vaccine | 3 doses tot | al | | X | X | X | | | | | | | |
| GM-CSF | 12 doses to | otal | | X (+3 days) | X<br>(+3<br>days) | X<br>(+3<br>days) | | | | | | | |

## > Treatment Group B: Lenalidomide and GM-CSF

If you are assigned to Treatment Group B, you will get: lenalidomide and GM-CSF injections.

You will take lenalidomide every day for 2 years or until your disease returns. You will receive the enough pills for 1 cycle (28 days in each cycle) at a time. It's important to take the pill at the same time every day. Be sure to talk with your doctor to figure out a good time to take the pill every day.

You will also get an injection of GM-CSF in upper thigh. You will get the GM-CSF injection every day for 4 days starting the first day of cycles 2, 3 and 4. This will either be given to you in the clinic or you will be taught to give the injections to yourself at home.

See **Table 3** for a timeline of the drugs for Treatment Group B.

**Table 3: Treatment Group B** 

| | | | Timeline for Maintenance Treatment Drugs | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group B<br>drugs: | Amount: | Cycle:<br>(28 days in<br>each cycle) | 1 | 2 | 3 | 4 | 6 | 9 | 12 | 15 | 18 | 21 | 24 |
| Lenalidomide | 1 dose every d | lay for 2 | X | X | X | X | X | X | X | X | X | X | X |
| GM-CSF | 12 doses total | | | X<br>(+ 3<br>days) | X<br>(+ 3<br>days) | X<br>(+ 3<br>days) | | | | | | | |

## > Treatment Group C: Lenalidomide

If you are assigned to Treatment Group C, you will take lenalidomide every day for 2 years or until your disease returns. You will receive enough pills for 1 cycle (28 days in each cycle) at a time. It's important to take the pill at the same time every day. Be sure to talk with your doctor to figure out a good time to take the pill every day.

## Maintenance treatment dose (All treatment groups)

#### How We Will Give You Lenalidomide

Lenalidomide is available only from a certified pharmacy through the Revlimid REMS® program. During maintenance therapy, only a 28-day supply (1 cycle) will be given to you at a time.

If this is the first time you've taken lenalidomide, you'll have to sign-up, or register, for the program. This will include a separate consent process, which calls out the reproductive risks of taking this medicine. You'll have to give your name, address, phone number, birth date, and social security number to sign-up for the program. This information will be provided to Celgene Corporation and Biologics Incorporated to show you're taking part in this study.

After you're registered, you'll be counseled at the site or through the program:

- When you're first given the drug
- At least every 28 days while you're taking it, and

• When you stop taking it

#### You will be counseled about:

- Side effects
- Not sharing lenalidomide (or other study drugs)
- Risks of exposing a fetus (unborn baby)
- Donating blood
- How to take the pills

We'll give you the, "Lenalidomide Information Sheet for Patients Enrolled in Clinical Research Studies" with each new supply of lenalidomide to remind you of these safety issues.

## How to Take the Lenalidomide Pills

- Swallow the whole lenalidomide pill with water at the same time each day. Do <u>not</u> break, chew or open the capsules.
- If you miss a dose, take it as soon as you remember on the same day. If you miss taking your dose for the entire day, take your regular dose the next scheduled day (do <u>not</u> take a double dose to make up for the missed dose).
- If you take more than the prescribed dose you should seek emergency medical care if needed and contact study staff right away.
- Women who can become pregnant that care for you <u>should wear gloves</u> whenever they need to touch the lenalidomide pills or bottles.

## **Checking Your Health**

We will watch your health closely during your maintenance treatment, including how well your organs work. We will lower your dose if your organs don't handle the treatment well.

We won't start a new cycle until your organs work well again. If we lower your dose and then your organs start working normally, we may raise your dose again.

We will stop the maintenance treatment if you:

• Have a serious side effect

- Have low blood cell counts
- Are a woman and become pregnant, or there is a chance that you are pregnant
- Go more than 56 days before starting a new maintenance treatment cycle
- Don't follow the study directions, or
- Choose to leave the study.

You will need to visit your clinic for several check-ups and tests during your maintenance treatment. These tests are shown in **Table 4. These assessments are standard of care for patients receiving lenalidomide maintenance therapy.** 

**Table 4. Timeline of Tests Before and During Your Maintenance Treatment** 

| Tests | Before<br>you're<br>Random | Ti | Timeline for Maintenance Treatment Tests (CYCLES) | | | | | | | Timeline for<br>Post-Transplant<br>Tests (Months) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | ized | 1 | 2 | 3 | 4 | 6 | 9 | 12 | 15 | 8 | 21 | 24 | 6T | 2T | 24T |
| Physical exam, height, and weight | X | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Tests for toxicities, and infections | X | X | X | X | X | X | X | | X | | X | X | | | |
| Blood tests for<br>cell counts,<br>liver and<br>kidney<br>function | X | X | X | X | X | X | X | X | X | X | X | X | | | |
| Tests to see<br>how much<br>cancer you<br>still have | X | | | X | | X | X | X | X | X | X | X | X | X | X |
| Pregnancy test<br>(women able<br>to have<br>children) | X | X | X | X | X | X | X | X | X | X | X | X | | | |

## **Blood and Bone Marrow Samples**

Throughout the study, we will collect blood and marrow samples to check if the treatments are working. These samples are being done as a part of the standard of care disease assessment. In addition, blood and marrow samples are also collected as part of this research study to check your immune response to the vaccine and are not part of your standard of care. The maximum amount of blood we will collect for this study in one day is 70mL (approximately 4.5 tablespoons). If more blood is required at a particular time, we will collect blood on 2 or more days spread out over 1-2 weeks.

The maximum amount of bone marrow sample we will collect is 37mL (approximately 2.5 tablespoons). **Table 5** shows the timeline and amount of samples we may collect from you during the study.

Table 5: Timeline and Sample Amount Collected during Study (in approximate tablespoons (Tbsp) or teaspoons (tsp))

| | When you join | Before | Maintenance Cycles | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Sample | the<br>study | you're<br>randomized | 1 | 2 | 2<br>(day 7) | 3 | 4 | 4<br>(day 7) | 9 |
| Bone marrow | 2.5 Tbsp | 1 tsp | | | | | | | 2 tsp |
| Optional bone<br>marrow<br>samples for<br>future research | <1 tsp | <1 tsp | | | | | | | <1 tsp |
| Blood-forming cells | 6.5 Tbsp<br>*over 10<br>days | 2 Tbsp | 4.5<br>Tbsp | 4.5<br>Tbsp | 4<br>Tbsp | 4.5<br>Tbsp | 4.5<br>Tbsp | 4 Tbsp | 4.5<br>Tbsp |
| Optional blood<br>samples for<br>future research | 1.5 tsp | 1.5 tsp | | | | | | | 1.5 tsp |

## 6. Risks and Discomforts

You may have side effects while on the study. Side effects can range from mild to serious. The risks and discomforts of autologous transplant are the same if you join this study, or if you don't join this study.

You might do better or worse than you would with a standard transplant. Your healthcare team may give you medicines to help with side effects like nausea (feeling sick to your stomach). In some cases, side effects can last a long time or may never go away.

### Risks of Making the Vaccine

We will collect bone marrow samples on all patients.

We will take the bone marrow samples from your hip bone with a large needle. This is called a bone marrow aspirate. After, you may feel pain and bleed at the site where the needle went in your hip. A small number of patients will have pain that runs down their legs, pain that lasts more than a few days, and/or get an infection.

If you are assigned to Treatment Group A, we will collect blood and bone marrow samples to make the vaccine (see **Table 5. Timeline and Sample Amount Collected during Study**).

We will also collect extra samples of blood through a catheter in your neck or chest (leukaphereis). The risks of leukapheresis include:

- Bleeding
- Punctured lung (hole in lung)
- Infection
- Low blood cell counts.

#### **Risks of Medications**

The risks of the chemotherapy and maintenance drugs you will get as part of the treatment are listed below.

# **Melphalan - Conditioning Regimen Drug (Before Transplant)**

| Likely (May happen in more than 20% of patients) | Less Likely (May happen in less than 20% of patients) | Rare, but Serious (May happen in less than 2% of patients) |
|---|---|---|
| <ul> <li>Loss of appetite</li> <li>Constipation</li> <li>Diarrhea</li> <li>Nausea (feeling sick to your stomach)</li> <li>Vomiting (throwing up)</li> <li>Temporary hair loss</li> <li>Sensitive skin</li> <li>Infection</li> <li>Low number of white blood cells</li> <li>Low number of platelets in the blood with increased risk of bleeding</li> <li>Anemia (low number of red blood cells)</li> <li>Mouth sores</li> <li>Sore throat (red with swelling)</li> <li>Skin breakdown (if drug leaks from vein)</li> </ul> | <ul> <li>Changes in heart beat</li> <li>Dizzy</li> <li>Feeling faint</li> <li>Shortness of breath</li> <li>Hepatitis (swelling of the liver)</li> <li>Kidney failure</li> <li>Weight loss</li> <li>Feeling weak</li> </ul> | <ul> <li>Allergic reaction</li> <li>Lung infection</li> <li>Scarring of lung tissue</li> <li>Seizure</li> <li>Vasculitis (inflammation of blood vessels)</li> <li>Low blood pressure</li> <li>Sweating too much</li> <li>Sterility (unable to have children)</li> <li>Liver damage</li> <li>Heart stops beating</li> <li>New cancer of bone marrow cells</li> </ul> |

# Vaccine

| Likely (May happen in more than 20% of patients) | Less Likely (May happen in less than 20% of patients) | Rare, but Serious (May happen in less than 2% of patients) |
|---|---|---|
| <ul> <li>Twitching injection site)</li> <li>Itching (general or at injection site)</li> <li>Discomfort (at injection site)</li> <li>Swelling (at injection site)</li> <li>Bruising at the injection site</li> </ul> | <ul> <li>Fluid retention (too much water in your body)</li> <li>Fatigue</li> <li>Muscle aches</li> <li>Itching</li> <li>Fever</li> <li>Abnormal Antinuclear Antibody (ANA) blood test</li> <li>Decreased white blood cell count (including neutrophils)</li> <li>Headache</li> <li>Diarrhea</li> <li>Feeling light headed</li> <li>Flu-like symptoms</li> <li>Night sweats</li> </ul> | <ul> <li>Allergic reaction leading to rashes, joint pain, kidney, heart or lung damage, drop in blood counts</li> <li>Tumor growth or the spread of your cancer</li> <li>Infection at the vaccine site</li> <li>Change in thyroid function (fatigue, weight gain, sensitivity to cold and lack of interest or emotion)</li> <li>Pulmonary embolus (blood clot in the lungs)</li> </ul> |

| Likely (May happen in more than 20% of patients) | Less Likely (May happen in less than 20% of patients) | Rare, but Serious (May happen in less than 2% of patients) |
|---|---|---|
| | <ul> <li>Elevated TSH (TSH is a thyroid hormone)</li> <li>Candida infection</li> </ul> | |

# **GM-CSF** (Leukine)

| Likely | Less Likely | Rare, but Serious |
|---|---|---|
| (May happen in more than 20% of patients) | (May happen in less than 20% of patients) | (May happen in less than 2% of patients) |
| • Fever | • Rapid, irregular heartbeats | Blood clots |
| • Chills | • Feeling lightheaded or dizzy | |
| • Nausea | | |
| Vomiting | Allergic reaction | |
| Diarrhea | • Fluid in lungs or around your heart | |
| • Fatigue | • Changes in vision | |
| Feeling weak | Low blood cell counts | |
| Headache | • Infection at needle | |
| Loss of appetite | injection site | |
| • Flushed face (red or pink cheeks) | | |
| Bone and muscle pain in arms, legs and feet | | |
| Red skin, swelling, or itching at needle injection site | | |
| Low blood pressure | | |
| Shortness of Breath | | |

# Lenalidomide- Maintenance Treatment Drug

| Likely | Less Likely | Rare, but Serious |
|---|---|---|
| (May happen in more than 10% of patients) | (May happen in less than 10% of patients) | (May happen in less than 2% of patients) |
| <ul> <li>Low number of white blood cells (with or without fever)</li> <li>Anemia; Decrease in cells that help your blood clot</li> <li>Vision Blurred</li> <li>Diarrhea</li> <li>Pain, Constipation</li> <li>Indigestion</li> <li>Nausea</li> <li>Vomiting</li> <li>Feeling weak and unwell</li> <li>Tired</li> <li>Swelling</li> <li>Fever</li> <li>Chills</li> <li>Pneumonia or other infections</li> <li>Sore throat</li> <li>Stuffy nose</li> <li>Weight loss</li> <li>Decreased appetite</li> <li>High blood sugar</li> </ul> | <ul> <li>Abnormally low number of blood cells</li> <li>Destruction of red blood cells</li> <li>Heart attack</li> <li>Abnormal heart beats</li> <li>Heart stops working</li> <li>Low oxygen to heart tissue</li> <li>Dry mouth</li> <li>Decreased action of intestine</li> <li>Bile flow from liver slowed or blocked</li> <li>Gout</li> <li>Fall</li> <li>Bruise</li> <li>Lowered level of consciousness with drowsiness, listlessness, and apathy</li> <li>Abnormal liver lab tests</li> <li>Increase in liver protein that indicates inflammation in body</li> <li>Loss of fluid</li> <li>Diabetes</li> <li>High uric acid in blood</li> <li>Iron build up in body</li> </ul> | <ul> <li>Swelling of lungs</li> <li>Over and underactive thyroid</li> <li>Severe allergic conditions including: Swelling under skin; Severe skin reactions involving lining of the nose, mouth, stomach and intestines or rash leading to the separation of the top layer of skin</li> <li>Tumor Lysis Syndrome (TLS) is caused by the sudden, rapid death of cancer cells in response to treatment. When cancer cells die they may spill their inner (intracellular) contents, which accumulate faster than they can be eliminated. This debris from the cancer cells can change the balance of the chemistry of the body, which can be dangerous.</li> </ul> |

- Chemical imbalance in blood
- Pain including muscles, joints, and non-cardiac chest pain
- Dizziness
- Altered sense of taste
- Headache
- Eye lens cloudy
- Abnormal sense of touch
- Pain and decreased sensation in nerves
- Shaking
- Cough
- Shortness of breath
- Nosebleed
- Blood clot in lower extremities, lungs, heart, brain, and other organs
- Dry skin
- Itching
- Allergic reaction
- Feeling sad
- Not sleeping well

- Muscle weakness
- Cancer
- Stroke
- Tingling of skin
- Fainting
- Moody
- Kidney failure
- Breathing disorder
- Excessive sweating
- Night sweats
- Skin redness
- Swelling of skin filled with blood
- Swelling of blood vessels
- High or low blood pressure
- Blood not getting to extremities
- Clot in vein
- Sudden increase in tumor size
- Rapid death of cancer cells where the accumulating contents of dying cancer cells cause an imbalance in the chemistry of the body which can lead to kidney damage
- Blood cancer that causes decreased number of red blood cells, white blood cells, and platelets because they do not develop normally.

You <u>shouldn't</u> donate blood while you're in the study and for 28 days after you stop taking lenalidomide.

#### Risk to the Unborn

Lenalidomide can cause <u>severe birth defects or death of a baby</u> if the mother or the father is taking this medicine at the time of conception or during pregnancy. **Because of this, it is extremely important that you don't get pregnant while you're taking lenalidomide.** 

If you're pregnant or nursing, you're not eligible to take part in this study. Women who can become pregnant must use <u>at least 2 forms of effective birth control</u> while in the study or abstain from all reproductive sexual intercourse. Effective birth control is defined as the following:

- 1. Refraining from all acts of vaginal sex (abstinence)
- 2. Consistent use of birth control pills
- 3. Injectable birth control methods (Depo-Provera, Norplant)
- 4. Tubal sterilization or male partner who has undergone a vasectomy
- 5. Placement of an IUD (intrauterine device)
- 6. Use of a cervical cap or a diaphragm with contraceptive jelly and/or condoms with contraceptive foam every time you have sex.

Females taking lenalidomide have blood clots more often. Because of this, you should talk to your doctor about birth control pills and hormone replacement therapy, and the risks and benefits.

You do not need to use effective birth control only if you are a woman and cannot have children because you:

- Had a hysterectomy (your ovaries and uterus were removed), OR
- Had a bilateral oophorectomy (your ovaries were removed), OR
- Went through menopause (post-menopausal).

#### Reproductive Risks

The drugs used in this research study may damage your reproductive organs, affect your ability to have children, or cause birth defects if you take them while you are pregnant or nursing.

Both women who can become pregnant <u>and</u> their male partners should use birth control while on this study and for 28 days after maintenance treatment is stopped. **If you or your partner** becomes pregnant during this study, you must tell the study doctor immediately.

Your doctor will discuss the risks to your unborn child and options with you.

It is important that females who aren't pregnant or nursing don't become pregnant while part of the study. If you are a woman and become pregnant while on this study, we will stop the maintenance treatment drug right away.

Your study doctor will watch your health closely while you are pregnant and for 30 days after the pregnancy ends.

#### Females who join the study

If you are female and can become pregnant, you will need to take a pregnancy test before you start the study. You should discuss ways to prevent pregnancy while you're in the study. Women who have gone through puberty might experience irregular menstrual cycles or their cycle might stop forever. This doesn't mean that you can't become pregnant. You must still use 2 effective forms of birth control during the study and continue with it for 28 days after you finish maintenance treatment.

Be sure to talk with your doctor about options for fertility planning, like storing your eggs, before starting chemotherapy treatment.

#### Males who join the study

If you are male, your body may not be able to produce sperm (become sterile). Be sure to talk with your doctor about options for fertility planning, like banking your sperm, before starting chemotherapy treatment.

#### Damage to the vital organs in your body

Your vital organs include your heart, lungs, liver, intestines, kidneys, bladder and brain. The chemotherapy drugs may hurt these organs. You may develop lung problems from chemotherapy or an infection.

Some patients can have veno-occlusive disease (VOD) of the liver. Patients with VOD become jaundiced (yellow skin), have problems with their liver, retain too much water (feel swollen and uncomfortable), and have stomach swelling and pain.

If there is serious damage to your vital organs, you may have to stay in the hospital longer or return to the hospital after your transplant. Many patients get better, but these complications can cause permanent damage to your organs or death.

#### Relapse (return) of disease or a new blood cancer

Your disease may come back even if the transplant was successful at first.

We don't know if new blood cancers are caused by lenalidomide or other drugs. Other research looked at the number of patients who got new blood cancers after taking lenalidomide for:

- Diseases other than multiple myeloma, AND
- Relapsed multiple myeloma.

In these studies, no difference was shown in the number of patients who got new blood cancers.

Researchers for other studies of lenalidomide are still watching patients to see if they get new blood cancers. We will give you any new information that we learn about new blood cancers.

#### All Patients Taking Lenalidomide

In order to participate in this study you must register into and follow the requirements of the REVLIMID REMS<sup>TM</sup> program of Celgene Corporation. This program provides education and counseling on the risks of fetal exposure, blood clots and reduced blood counts. You will be required to receive counseling every 28 days during treatment with lenalidomide, follow the pregnancy testing and birth control requirements of the program that are appropriate for you and take telephone surveys regarding your compliance with the program.

You have been informed of the risk of birth defects. If you are female, you agree not to become pregnant while taking lenalidomide. For this reason, lenalidomide is provided to patients under a special distribution program called REVLIMID REMS TM.

#### Other Information:

There may be some unknown or unanticipated discomforts or risks associated with this treatment in addition to those specified above, but every precaution will be taken to assure your personal safety and to minimize discomforts.

Throughout the study, the researchers will tell you of new information that might affect your decision to remain in the study.

If you wish to discuss the information above or any other discomforts you may experience, you may ask questions now or call your doctor \_\_\_\_\_\_\_, the Principal Investigator or contact person listed on the front page of this form.

#### **Other Risks**

#### Serious infections

It may take many months for your immune system to recover from the chemotherapy and maintenance therapy drugs. There is an increased risk of infection during this time when your body is healing. We will give you drugs to reduce the chance of infection, but they may not work. If you have an infection, you may have to stay in the hospital longer or return to the hospital after transplant. Many patients get better, but some infections can cause death.

#### Unforeseen Risks

Chemo drugs can damage your blood cells, which may cause a new blood cancer to grow. We know from other MM research studies, that more patients had a second cancer after chemo and/or autologous transplant with maintenance lenalidomide than those who didn't get lenalidomide. We don't know if taking lenalidomide for a long time raises the risk of having a second cancer.

Other new risks might appear at any time during the study. These risks might be different from what is listed in this Consent Form. There may be some unknown or unanticipated discomforts or risks associated with this treatment in addition to those specified above, but every precaution will be taken to assure your personal safety and to minimize discomforts.

## Other Treatments or Medicines

Some medicines react with each other, and it is important that you tell the study doctor or staff about any other drugs, treatments, or medicines you are taking. This includes non-prescription or over-the-counter medicines, vitamins, and herbal treatments.

It is also important that you tell the study staff about any changes to your medicines while you're in the study.

For more information about risks and side effects, ask your study doctor.

#### 7. Other Treatments

Participation in this study is optional. If you choose not to take part, you may still receive non-transplant treatments or an autologous or an allogeneic transplant to treat your disease. The treatment and evaluations you would receive could be very similar to what would receive if you join this study.

Your study doctor will talk with you about your options. If you decide not to participate in this study, your medical care will not be affected in any way.

Your other options may include:

- Treatment with other drugs, radiation, or a combination of drugs and radiation without a transplant.
- An allogeneic (donor) blood or marrow transplant that is not part of the study, or another type of transplant
- Participation in another clinical trial, if available (check with your doctor)
- No treatment for your blood cancer at this time
- Comfort care

Every treatment option has benefits and risks. Talk with your doctor about your treatment choices before you decide if you will take part in this study.

#### 8. Possible Benefits

Taking part in this study may or may not make your health better. The information from this study will help doctors learn more about drugs used to treat MM.

This information could help people with multiple myeloma who may need a transplant in the future.

## 9. New Information Available During the Study

During this research study, the study doctors may learn about new information about the study drugs or the risks and benefits of the study. If this happens, they will tell you about the new information. The new information may mean that you can no longer participate in the study, or that you may not want to continue in the study.

If this happens, the study doctor will stop your participation in the study and will offer you all available care to suit your needs and medical conditions.

# 10. Privacy, Confidentiality and Use of Information

Your privacy is very important to us. The study doctors will make every effort to protect it. The study doctors have a privacy permit to help protect your records if there is a court case. However, some of your medical information may be given out if required by law. If this should happen, the study doctors will do their best to make sure that any information that goes out to others will not identify who you are.

Data regarding your clinical situation, including follow-up after 2 years, may be obtained from the CIBMTR, which captures information on all US transplants.

All your medical and demographic information (such as race and ethnicity, gender and household income) will be kept private and confidential. (*Name of Transplant Center*) and the organizations listed below will not disclose your participation by any means of communication to any person or organization, except by your written request, or permission, or unless required by federal, state or local laws, or regulatory agencies.

The individuals below will have access to your research and medical information. They may use this information for inspections or audits to study the outcomes of your treatment. By agreeing to participate, you consent to such inspections and to the copying of parts of your records, if required by these organizations.

We may give out your personal information if required by law. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used.

Information about your transplant from your original medical records may be seen or sent to national and international transplant registries, including:

#### 1. /Institution/

- 2. The Center for International Blood and Marrow Transplant Research (CIBMTR)
- 3. The National Marrow Donor Program (NMDP)
- 4. The Food and Drug Administration (FDA)
- 5. The National Institutes of Health (NIH), which include the National Heart, Lung, and Blood Institute (NHLBI) and the National Cancer Institute (NCI)
- 6. Data and Coordinating Center of the Blood and Marrow Transplant Clinical Trials Network (BMT CTN)
- 7. Data and Safety Monitoring Board (DSMB), not part of /Institution/
- 8. Study investigators.
- 9. Celgene, the manufacturer of lenalidomide

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time. For questions about access to your medical records, please contact <a href="https://name/">name/</a> at <a href="https://name/">number</a>.

# 11. Ending Your Participation

The study doctor or the study sponsor may stop the study at any time, and we may ask you to leave the study. We may ask you to leave the study if you do not follow directions or if you suffer from side effects of the treatment. If we ask you to leave the study, the reasons will be discussed with you. Possible reasons to end your participation in this study include:

- 1. You do not meet the study requirements.
- 2. You need a medical treatment not allowed in this study.
- 3. The study doctor decides that it would be harmful to you to stay in the study.

- 4. You are having serious side effects.
- 5. You become pregnant.
- 6. You cannot keep appointments or take study drugs as directed.
- 7. The study is stopped for any reason.

You could have serious health risks if you stop treatment during the conditioning process before you receive your transplant. If you stop taking the immune suppressing drugs (see **Section 6: Risks and Discomforts**) too soon after transplant, your body could reject the stem cells or you could develop serious complications and possibly die.

We ask that you talk with the research doctor and your regular doctor before you leave the study. Your doctors will tell you how to stop safely and talk with you about other treatment choices.

If you decide to leave this study after getting the study treatment, or are asked to leave by your doctor for medical reasons, you will need to come back to the doctor's office for tests for your safety. Even if you leave the study, the information collected from your participation will be included in the study evaluation, unless you specifically ask that it not be included.

| 12. | Physical Injury as a | Result of Participation | |
|---|---|---|---|
| It is in | portant that you tell your doc | etor,[investigator's n | name(s)] or study |
| staff if | you feel that you have been i | injured because of taking part in this study. | You can tell the |
| doctor | in person or call him/her at _ | [telephone number]. | |

You will get all available medical treatment if you are injured from taking part in this study. You and/or your health plan will be charged for this treatment. There is no provision for free medical care or monetary compensation from the study sponsor, The National Institutes of Health or the study contributor, Celgene Corporation.

In case you are injured in this study, you do not lose any of your legal rights to ask for or receive payment by signing this form.

# 13. Compensation or Payment

You will not be paid for your participation in this research study. You will not get compensation or reimbursement for any extra expenses (travel, meals, etc.) you may have through your participation on this trial.

Taking part in this study might help researchers make products to sell. Celgene or others may profit from these products. You will not have any rights to the patents or discoveries that could happen from this research, and you will not receive any payments from it.

#### 14. Costs and Reimbursements

Most of the visits for this research study are standard medical care for your autologous transplant and will be billed to your insurance company. You and/or your health plan/insurance company will need to pay for some or all of the costs of standard treatment in this study.

You or your insurance will <u>not</u> be charged for blood and marrow samples for research on this study. You will not pay for any extra tests that are being done for the study. Lenalidomide will be provided to you for free for two years. After that your doctor will discuss what treatment is best for you.

Some health plans will not pay these costs for people taking part in studies. Check with your health plan or insurance company to find out if they will pay.

For questions about your costs, financial responsibilities, and/or medical insurance coverage for your transplant and this study, please contact /Center/ Financial Counselor at /Number/.

For more information on clinical trials and insurance coverage, you can visit the National Cancer Institute's Web site at <a href="http://cancer.gov/clinicaltrials/understanding/insurance-coverage">http://cancer.gov/clinicaltrials/understanding/insurance-coverage</a>. You can print a copy of the "Clinical Trials and Insurance Coverage" information from this Web site.

Another way to get the information is to call 1-800-4-CANCER (1-800-422-6237) and ask them to send you a free copy.

#### 15. For More Information

If you need more information about this study, or if you have problems while taking part in this study, you can contact the study doctor or his/her staff.

They can be reached at the telephone numbers listed here:

[Insert name and contact details]

# 16. Contact Someone about Your Rights

If you wish to speak to someone not directly involved in the study, or if you have any complaints about any aspect of the project, the way it is being conducted or any questions about your rights as a research participant, then you may contact:

[Insert appropriate contact details]

The ethical aspects of this study have been reviewed and approved by *[name of IRB]*.

# 17. Blood and Bone Marrow Samples for Future Research (Optional)

This section of the informed consent form is about future research studies that will use blood and bone marrow samples from people who are taking part in the main study. You may choose to give samples for these future research studies if you want to. You can still be a part of the main study even if you say 'no' to give samples for future research studies.

Researchers are trying to learn more about how the human body processes the drugs used for transplant and how the body recovers after transplant. This research is meant to gain knowledge that may help people in the future and make transplants even more successful.

If you agree to provide blood and bone marrow samples, here is what will happen:

- We will collect 3 extra blood samples at the same time you have routine blood tests done (Table 3):
  - o Around the time of your enrollment
  - o About 2 months after your transplant
  - o Before the start of your 9<sup>th</sup> cycle of maintenance therapy
- The amount of blood collected from you is about 1 teaspoon (6 ml) each time.
- We will collect 3 bone marrow samples at the same time you have routine bone biopsies done. The amount of tissue collected from you is about a half of a teaspoon (3 mL) each time. We will collect samples at 3 different dates in the study (see **Table 3**):
  - o Around the time of your enrollment
  - o About 2 months after your transplant
  - o Before the start of your 9<sup>th</sup> cycle of maintenance therapy.
- The blood and bone marrow samples will be sent to the BMT CTN Repository for processing and storage. A repository is a place that protects, stores and sends out samples for approved research studies. All research samples will be given a bar code that cannot be linked to you by future researchers testing your samples.
- Materials stored in the Repository will be used mainly by clinicians and researchers in the BMT CTN network. In the future, the unused research samples and clinical data will be made available outside of this network.

- Researchers can apply to study the materials stored in the Repository. The BMT CTN Steering Committee and/or the BMT CTN Executive Committee must approve each request before they will share samples or information with researchers. This is to make sure that the investigators requesting the samples are qualified, and that the research is of high quality.
- DNA from your stored blood samples might be used in genome-wide association (GWA) studies for a future project either done or supported by the National Institutes of Health (NIH).
   Genome-wide association studies are a way for scientists to find genes that have a role in human disease or treatment. Each study can look at hundreds of thousands of genetic changes at the same time.

If your coded samples are used in such a study, the researcher is required to add your test results and sample information into a shared, public research database. This public database is called the NIH Genotype and Phenotype Database and it is managed by the National Center for Biotechnology Information (NCBI). The NCBI will never have any information that would identify you, or link you to your information or research samples.

Some general things you should know about letting us store your blood samples for research are:

- 1. We will only store samples from people who give us permission.
- 2. Research is meant to gain knowledge that my help people in the future. You will not get any direct benefit from taking part. Additionally, you or your doctor will not be given results and they will not be added to your medical record.
- 3. A possible risk is the loss of confidentiality about your medical information. We will use safety measures with both your samples and clinical information to make sure that your personal information will be kept private. The chance that this information will be given to someone else is extremely small.
- 4. Your blood will be used only for research and will not be sold. The research done with your blood may help to develop new products in the future. You will not get paid for any samples or for any products that may be developed from current or future research.

You can change your mind at any time about allowing us to use your samples and health information for research.

We ask that you contact [*Principal Investigator*] in writing and let him/her know you do not want us to use your research samples or health information for research. His/her mailing address is on the first page of this form. However, samples and information that have already been shared with other researchers cannot be taken back or destroyed.

## **Making Your Choice**

Please read each sentence below and think about your choice. After reading each sentence, please indicate your choice below. If you have any questions, please talk to your doctor or nurse, or call our research review board at [contact information].

No matter what you decide to do, it will not affect your care.

# **Statement of Consent for Research Samples**

The purpose of storing blood and tissue samples, the procedures involved, and the risks and benefits have been explained to me. I have asked all the questions I have at this time and I have been told whom to contact if I have more questions. I have been told that I will be given a signed copy of this consent form to keep.

I understand that I do not have to allow the use of my blood and tissue for research. If I decide to not let you store research samples now or in the future, it will not affect my medical care in any way.

I voluntarily agree that my blood, tissue, and information can be stored indefinitely by the BMT CTN and/or NHLBI Repositories for research to learn about, prevent, or treat health problems. I also understand that my DNA and health information may or may not be used in genome-wide association studies.

| Blood | |
|---|---|
| | I agree to allow my blood samples to be stored for research. |
| | I do not agree to allow my blood samples to be stored for research. |
| Во | ne marrow |
| | I agree to allow my bone marrow samples to be stored for research. |
| | I do not agree to allow my bone marrow samples to be stored for research. |
| Sig | nature Date |

Health Insurance Portability and Accountability Act 1 (HIPAA1) Authorization to use and disclose individual health information for research purpose

#### • Purpose:

As a research participant, I authorize the Principal Investigators and the researcher's staff to use and disclose my individual health information for the purpose of conducting the research study:

Phase II Multicenter Trial of Single Autologous Hematopoietic Cell Transplant Followed by Lenalidomide Maintenance for Multiple Myeloma with or without Vaccination with Dendritic Cell /Myeloma Fusions

• Individual Health Information to be Used or Disclosed:

My individual health information that may be used or disclosed to do this research includes:

- 1. Demographic information (for example, date of birth, sex, weight)
- 2. Medical history (for example, diagnosis, complications with prior treatment)
- 3. Findings from physical exams
- 4. Laboratory test results obtained at the time of work up and after transplant (for example, blood tests, biopsy results)
  - Parties Who May Disclose My Individual Health Information:

The researcher and the researcher's staff may collect my individual health information from:

[List hospitals, clinics or providers from which health care information can be requested]

• Parties Who May Receive or Use My Individual Health Information:

The individual health information disclosed by parties listed in item c and information disclosed by me during the course of the research may be received and used by the following parties:

- 1. Dr. David Avigan, Co-Principal Investigator
- 2. Dr. Nina Shah, Co-Principal Investigator
- 3. Dr. David Chung, Co-Principal Investigator

<sup>1</sup> HIPAA is the Health Insurance Portability and Accountability Act of 1996, a federal law related to privacy of health information

- 4. Celgene, its collaborators or designees
- 5. National Heart, Lung, and Blood Institute (NHLBI) and the National Cancer Institute (NCI), both of the National Institutes of Health (NIH),
- 6. Blood and Marrow Transplant Clinical Trials Network (BMT CTN) Data and Coordinating Center
- 7. <u>U.S. government agencies that are responsible for overseeing research</u> such as the Food and Drug Administration (FDA) and the Office of Human Research Protections (OHRP)
- 8. <u>U.S. government agencies that are responsible for overseeing public health concerns</u> such as the Centers for Disease Control (CDC) and federal, state and local health departments.

## • Right to Refuse to Sign this Authorization:

I do not have to sign this Authorization. If I decide not to sign the Authorization, I will not be allowed to participate in this study or receive any treatment related to research that is provided through the study.

My decision not to sign this authorization will not affect any other treatment, payment, or enrollment in health plans or eligibility for benefits.

## • Right to Revoke:

I can change my mind and withdraw this authorization at any time by sending a written notice to the Principal Investigator to inform the researcher of my decision.

If I withdraw this authorization, the researcher may only use and disclose the protected health information already collected for this research study. No further health information about me will be collected by or disclosed to the researcher for this study.

#### • Potential for Re-disclosure:

My individual health information disclosed under this authorization may be subject to redisclosure outside the research study and no longer protected.

Examples include potential disclosures for law enforcement purposes, mandated reporting or abuse or neglect, judicial proceedings, health oversight activities and public health measures.

#### • Genetic Information Nondiscrimination Act (GINA)

A new federal law (2009), called the Genetic Information Nondiscrimination Act (GINA) generally makes it illegal for health insurance companies, group health plans, and employers of 15 or more persons to discriminate against you based on your genetic information.

Health insurance companies and group health plans may not request your genetic information that we get from this research. This means that they must not use your genetic information when making decisions regarding insurability. Be aware that this new federal law will not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance.

• This authorization does not have an expiration date.

TITLE: Phase II Multicenter Trial of Single Autologous Hematopoietic Cell Transplant Followed by Lenalidomide Maintenance for Multiple Myeloma with or without Vaccination with Dendritic Cell /Myeloma Fusions

| PROTOCOL NUMBER: BMT CTN #1401 | | | |
|---|---|--|--|
| PRINCIPAL INVESTIGATOR: | | | |
| Name: Address: | | | |
| Phone: | | | |
| Fax: | | | |
| <ul> <li>I have read and understood this Consent Form. The nature and purposen explained to me.</li> <li>I have had the chance to ask questions, and understand the understand that I may ask questions at any time during the stud</li> </ul> | answers I have been given. I | | |
| • I freely agree to be a participant in the study. | | | |
| I understand that I may not directly benefit from taking part in the study. | | | |
| I understand that, while information gained during the study may be published, I will not be identified and my personal results will stay confidential. | | | |
| • I have had the chance to discuss my participation in this research or friend. | ch study with a family member | | |
| • I understand that I can leave this study at any time, and doing so or prevent me from receiving future treatment. | will not affect my current care | | |
| • I understand that I will be given a copy of this signed consent for | orm. | | |
| Participant Name | Date | | |
| Signature | Date | | |
| I certify that I have provided a verbal explanation of the details of the procedures and risks. I believe the participant has understood the | • | | |
| Name of Counseling Physician | Date | | |
| Signature of Counseling Physician | - Date | | |
| Ì | Q) | 1/ | 1 | r | C | T | 17 | V | T | CA | li | T | T | R | $I \Delta$ | I | 5 | 4 | λ | F | T | 'IA | 17 | 0 | R | k | 7 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| , | )/ | V | | , | | 11 | • | ν. | ,, | | | | ,,, | ١. | <i>1</i> / 1 | • | / L ] | | / V | 12 | , | v | , | • | /\ | 7 | |

# INFORMED CONSENT DOCUMENTS FOR BMT CTN 1401 OPTIONAL CORRELATIVE LABORATORY STUDY PARTICIPATION

#### **Informed Consent to Participate in Research**

Optional Correlative Laboratory Study Participation for patients enrolled on BMT CTN 1401 entitled "Phase II Multicenter Trial of Single Autologous Hematopoietic Cell Transplant Followed by Lenalidomide Maintenance for Multiple Myeloma with or without Vaccination with Dendritic Cell /Myeloma Fusions"

**Study Title:** Optional Correlative Laboratory Study Participation for patients enrolled on

BMT CTN 1401 "Phase II Multicenter Trial of Single Autologous Hematopoietic Cell Transplant Followed by Lenalidomide Maintenance for Multiple Myeloma with or without Vaccination with Dendritic Cell

/Myeloma Fusions"

Parent Study Title: Phase II Multicenter Trial of Single Autologous Hematopoietic Cell

Transplant Followed by Lenalidomide Maintenance for Multiple Myeloma

with or without Vaccination with Dendritic Cell /Myeloma Fusions

**Protocol:** BMT CTN 1401 v4.0

**Principal** 

**Investigator: Insert local PI information** 

**Sponsor:** The National Institutes of Health (NIH) is sponsoring this study by

providing financial support for the coordination of this study through the

Blood and Marrow Transplant Clinical Trials Network (BMT CTN).

## 1. Introduction

We invite you to participate in one or both of the optional correlative laboratory studies associated with the BMT CTN 1401 trial. You're being asked to join these optional studies because you were enrolled on BMT CTN 1401 and are being evaluated for randomization. Participation in these studies will involve you agreeing to allow investigators to either use previously collected research samples required by the primary trial and/or provide additional blood and marrow samples during your participation on the primary BMT CTN 1401 trial.

It is your choice to participate in these optional studies and to provide additional blood or bone marrow samples for this optional research. Even if you decide not to participate in these optional research studies, you can still participate on the primary BMT CTN 1401 study.

This Consent Form will tell you about the purpose of the optional research studies, the clinical samples needed for this research, the possible risks and benefits, other options available to you, and your rights as a research participant.

Everyone who takes part in research at [insert facility name] should know that:

- Being in any research study is voluntary.
- You will not directly benefit from being in the study. Knowledge we gain from this study may benefit others.
- If you give blood and bone marrow samples for research, you can change your mind at any time. The blood and marrow samples that you already provided will be used for research but no further research will be done after you change your mind.
- If you decide to quit the study, it will not affect your at [insert name of facility or institution].
- Please ask the study staff questions about anything that you do not understand, or if you would like to have more information.
- You can ask questions now or any time during the study.
- Please take the time you need to talk about the study with your doctor, study staff, and your family and friends. It is your decision to provide samples for research. If you decide to join, please sign and date the end of the Consent Form.

# 2. Study Background

The National Institutes of Health (NIH), through the Blood and Marrow Transplant Clinical Trials Network (BMT CTN), are providing staff support and money for this research study. The BMT CTN and the NIH will make decisions about how to manage the study.

For participation in one or both of these optional research studies, you will be asked to provide blood or bone marrow samples that will be shipped to a lab for further testing. Your doctor will discuss the research studies that are available to you as a part of this study.

## 3. Study Purpose

We are conducting these additional laboratory studies to further our understanding and knowledge about how the treatments you receive as part of the parent study (BMT CTN 1401) work.

## 4. Rights to Ask Questions and/or Withdraw

You have the right to ask questions about the study at any time. If you have questions about your rights as a participant or you want to leave the study, please contact:

#### [insert contact info]

Participating in either of these optional research studies is voluntary. You can choose not to be in these studies or leave either study at any time. However, some of the blood and bone marrow already donated may have already been used for research. If you choose not to take part or leave one of these studies, it will not affect your regular medical care in any way.

Your study doctor and study staff will be available to answer any questions that you may have about taking part in or leaving these optional research studies.

# 5. Study Treatment and Tests

There are two different research studies associated with the primary parent trial (BMT CTN 1401) that you are participating in. You doctor will explain which studies you are being asked to participate on at the end of this consent form and you will be presented with one or two more informed consent forms. These consent forms will go over the study tests in detail. The schedule of blood or bone marrow collections will depend on which studies you agree to participate in. If you would like to participate in this optional research, you will be asked to sign this informed consent form along with the other consent form(s) associated with the optional research your doctor is asking you to be a part of.

If you agree to participate on either of these research studies, your blood and or bone marrow will be shipped to laboratories at either Beth Israel Deaconess Medical Center and/or the University of Wisconsin. All research samples will be given a bar coded ID that cannot be linked to you by the researchers testing your samples. Samples will not be used for purposes other than those specified in this consent form

#### 6. Risks and Discomforts

Information about your demographics, disease, and response to the treatments you receive as part of the main clinical study may be provided to the investigators listed in the privacy portion of this consent form. This information is used to help the investigators understand how the research samples correlate to your disease. There are no major risks to having your blood or bone marrow drawn. It can be uncomfortable to have your blood and bone marrow taken and it can sometimes leave a bruise. You might faint, but this is unlikely to happen. Only trained people will take your blood and bone marrow

A possible risk is the loss of confidentiality about your medical information. We will use safety measures with both your samples and clinical information to make sure that your personal information will be kept private. The chance that this information will be given to someone else is extremely small.

For more information about risks and side effects, ask your study doctor.

#### 7. Other Treatments

Participation in this study is optional. The alternative to participating on this research sample study, is not agreeing to provide blood or bone marrow samples. If you choose not to take part, your treatment on BMT CTN 1401 will not be affected

This information could help people with multiple myeloma who may need a transplant in the future

#### 8. Possible Benefits

Taking part in this study will not make your health better. You will not get any direct benefit from taking part in this study. The information from this study will help doctors and researchers learn more about how well unrelated transplant works as treatment for people with a blood disease.

# 9. Privacy, Confidentiality and Use of Information

Your privacy is very important to us. The study doctors will make every effort to protect it. The study doctors have a privacy permit to help protect your records if there is a court case. However, some of your medical information may be given out if required by law. If this should happen, the study doctors will do their best to make sure that any information that goes out to others will not identify who you are.

Data regarding your clinical situation, including follow-up after 2 years, may be obtained from the CIBMTR, which captures information on all US transplants.

All your medical and demographic information (such as race and ethnicity, gender and household income) will be kept private and confidential. (Name of Transplant Center) and the organizations listed below will not disclose your participation by any means of communication to any person or

organization, except by your written request, or permission, or unless required by federal, state or local laws, or regulatory agencies.

The individuals below will have access to your research and medical information. They may use this information for inspections or audits to study the outcomes of your treatment. By agreeing to participate, you consent to such inspections and to the copying of parts of your records, if required by these organizations.

We may give out your personal information if required by law. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used.

Information about your transplant, research samples, and treatment on BMT CTN 1401 from your original medical records may be seen or sent to national and international transplant registries, including:

#### 1. /Institution/

- 2. The Center for International Blood and Marrow Transplant Research (CIBMTR)
- 3. The National Marrow Donor Program (NMDP)
- 4. The Food and Drug Administration (FDA)
- 5. The National Institutes of Health (NIH), which include the National Heart, Lung, and Blood Institute (NHLBI) and the National Cancer Institute (NCI)
- 6. Data and Coordinating Center of the Blood and Marrow Transplant Clinical Trials Network (BMT CTN)
- 7. Data and Safety Monitoring Board (DSMB), not part of /Institution/
- 8. Study investigators.
- 9. Dr. David Avigan and laboratory staff at Beth Israel Deaconess Medical Center/Dana Farber Cancer Institute
- 10. Dr. Fotis Asimakopoulos and laboratory staff at University of Wisconsin and at Medical College of Wisconsin.
- 11. Celgene, the manufacturer of lenalidomide

DNA from your blood samples might be used in genome-wide association (GWA) studies for a future project either done or supported by the National Institutes of Health (NIH). Genome-wide

association studies are a way for scientists to find genes that have a role in human disease or treatment. Each study can look at hundreds of thousands of genetic changes at the same time.

If your coded samples are used in such a study, the researcher is required to add your test results and sample information into a shared, public research database. This public database is called the NIH Genotype and Phenotype Database and it is managed by the National Center for Biotechnology Information (NCBI). The NCBI will never have any information that would identify you, or link you to your information or research samples.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

For questions about access to your medical records, please contact /name/ at /number.

## 10. Ending Your Participation

The study doctor or the study sponsor may stop the study at any time, and we may ask you to leave the study. We may ask you to leave the study if you do not follow directions or if you suffer from side effects of the treatment. If we ask you to leave the study, the reasons will be discussed with you. Possible reasons to end your participation in this study include:

- 1. You do not meet the study requirements.
- 2. The study doctor decides that it would be harmful to you to stay in the study.
- 3. You become unable to donate blood or bone marrow for any reason
- 4. The study is stopped for any reason.

Even if you leave the study, the information collected from your participation will be included in the study evaluation, unless you specifically ask that it not be included.

| 11. Physical Injury as a Result of Participation | |
|---|---|
| It is important that you tell your doctor, | _[investigator's name(s)] or study |
| staff if you feel that you have been injured because of taking p | part in this study. You can tell the |
| doctor in person or call him/her at [telep | phone number]. |

You will get all available medical treatment if you are injured from taking part in this study. You and/or your health plan will be charged for this treatment. There is no provision for free medical care or monetary compensation from the study sponsor, The National Institutes of Health or the study contributor, Celgene Corporation.

In case you are injured in this study, you do not lose any of your legal rights to ask for or receive payment by signing this form.

## 12. Payment and Study Costs

You will not be paid for donating your blood and/or bone marrow. You will not be paid or reimbursed for any extra expenses (travel, meals, etc.) you may have to donate blood and bone marrow.

Your blood and marrow will be used only for research and will not be sold. The research done with your blood may help to develop new products in the future. You will not get paid for any samples or for any products that may be developed from current or future research.

The visits for this research study are standard medical care for your autologous transplant and will be billed to your insurance company. You and/or your health plan/insurance company will need to pay for some or all of the costs of standard treatment in this study.

For questions about your costs, financial responsibilities, and/or medical insurance coverage for your transplant and this study, please contact /Center/ Financial Counselor at /Number/.

#### 13. For More Information

If you need more information about these studies, or if you have problems while taking part in either of these studies, you can contact the study doctor or his/her staff.

They can be reached at the telephone numbers listed here:

[Insert name and contact details]

# 14. Contact Someone about Your Rights

If you wish to speak to someone not directly involved in the study, or if you have any complaints about any aspect of the project, the way it is being conducted or any questions about your rights as a research participant, then you may contact:

## [Insert appropriate contact details]

The ethical aspects of this study have been reviewed and approved by *[name of IRB]*.

Health Insurance Portability and Accountability Act 1 (HIPAA2) Authorization to use and disclose individual health information for research purpose

<sup>2</sup> HIPAA is the Health Insurance Portability and Accountability Act of 1996, a federal law related to privacy of health information

#### • Purpose:

As a research participant, I authorize the Principal Investigators and the researcher's staff to use and disclose my individual health information for the purpose of conducting either of the research studies described in this consent:

Optional Correlative Laboratory Study Participation for patients enrolled on "Phase II

Multicenter Trial of Single Autologous Hematopoietic Cell Transplant Followed by

Lenalidomide Maintenance for Multiple Myeloma with or without Vaccination with Dendritic

Cell /Myeloma Fusions"

#### • Individual Health Information to be Used or Disclosed:

My individual health information that may be used or disclosed to do this research includes:

- 1. Demographic information (for example, date of birth, sex, weight)
- 2. Medical history (for example, diagnosis, complications with prior treatment)
- 3. Findings from physical exams
- 4. Laboratory test results obtained at the time of work up and after transplant (for example, blood tests, biopsy results)

#### • Parties Who May Disclose My Individual Health Information:

The researcher and the researcher's staff may collect my individual health information from:

[List hospitals, clinics or providers from which health care information can be requested].

#### • Parties Who May Receive or Use My Individual Health Information:

The individual health information disclosed by parties listed in item c and information disclosed by me during the course of the research may be received and used by the following parties:

- 1. Dr. David Avigan, Co-Principal Investigator
- 2. Dr. Nina Shah, Co-Principal Investigator
- 3. Dr. David Chung, Co-Principal Investigator
- 4. Laboratory staff at Beth Israel Deaconess Medical Center/Dana Farber Cancer Institute
- 5. Dr. Fotis Asimakopoulos and laboratory staff at University of Wisconsin and at Medical College of Wisconsin.

- 6. Celgene, its collaborators or designees
- 7. National Heart, Lung, and Blood Institute (NHLBI) and the National Cancer Institute (NCI), both of the National Institutes of Health (NIH),
- 8. Blood and Marrow Transplant Clinical Trials Network (BMT CTN) Data and Coordinating Center
- 9. <u>U.S. government agencies that are responsible for overseeing research</u> such as the Food and Drug Administration (FDA) and the Office of Human Research Protections (OHRP)
- 10. <u>U.S.</u> government agencies that are responsible for overseeing public health concerns such as the Centers for Disease Control (CDC) and federal, state and local health departments.

#### • Right to Refuse to Sign this Authorization:

I do not have to sign this Authorization. If I decide not to sign the Authorization, I will not be allowed to participate in this study.

My decision not to sign this authorization will not affect any other treatment, payment, or enrollment in health plans or eligibility for benefits.

#### • Right to Revoke:

I can change my mind and withdraw this authorization at any time by sending a written notice to the Principal Investigator to inform the researcher of my decision.

If I withdraw this authorization, the researcher may only use and disclose the protected health information already collected for this research study. No further health information about me will be collected by or disclosed to the researcher for this study.

#### • Potential for Re-disclosure:

My individual health information disclosed under this authorization may be subject to redisclosure outside the research study and no longer protected.

Examples include potential disclosures for law enforcement purposes, mandated reporting or abuse or neglect, judicial proceedings, health oversight activities and public health measures.

#### • Genetic Information Nondiscrimination Act (GINA)

A federal law (2009), called the Genetic Information Nondiscrimination Act (GINA) generally makes it illegal for health insurance companies, group health plans, and employers of 15 or more persons to discriminate against you based on your genetic information.

Health insurance companies and group health plans may not request your genetic information that we get from this research. This means that they must not use your genetic information when making decisions regarding insurability. Be aware that this federal law will not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance.

• This authorization does not have an expiration date.

TITLE: Optional Correlative Laboratory Study Participation for Patients Enrolled on BMT CTN 1401 entitled, "Phase II Multicenter Trial of Single Autologous Hematopoietic Cell Transplant Followed by Lenalidomide Maintenance for Multiple Myeloma with or without Vaccination with Dendritic Cell /Myeloma Fusions"

| PROTOCOL NUMBER: BMT CTN #1401 PRINCIPAL INVESTIGATOR: Name: Address: Email: Phone: Fax: | |
|---|---|
| <ul> <li>I have read and understood this Consent Form. The nature and purp been explained to me.</li> <li>I have had the chance to ask questions, and understand the at understand that I may ask questions at any time during the study.</li> </ul> | nswers I have been given. |
| • I freely agree to be a participant in the study. | |
| • I understand that I may not directly benefit from taking part in the | e study. |
| • I understand that, while information gained during the study maidentified and my personal results will stay confidential. | y be published, I will not be |
| • I have had the chance to discuss my participation in this research or friend. | study with a family member |
| • I understand that I can leave this study at any time, and doing so will not affect my current or prevent me from receiving future treatment. | |
| • I understand that I will be given a copy of this signed consent for | rm. |
| Participant Name | Date |
| Signature | Date |

| I certify that I have provided a verbal explanation of the details of the research study, includi the procedures and risks. I believe the participant has understood the information provided. | |
|---|---|
| Name of Counseling Physician | Date |
| Signature of Counseling Physician | Date |

### **Supplemental Informed Consent Form to Participate in Research**

**Study Title:** Characterization of the T cell immune response and myeloma genomic signature as predictors of immunologic and clinical response

**Parent Study Title:** Phase II Multicenter Trial of Single Autologous Hematopoietic Cell Transplant Followed by Lenalidomide Maintenance for Multiple Myeloma with or without Vaccination with Dendritic Cell /Myeloma Fusions

#### A. What is this Document?

The purpose of this document is to give you more information on the specific research sample study your physician is asking for your consent to join. This document will explain further details of what samples are collected, why they are being collected, and where they are being sent. Details about risks, study participation, and your rights are explained in the primary informed consent form that your doctor already presented to you.

## B. Why am I here?

You are being asked to participate in this study because you are participating on BMT CTN 1401 and are approaching the randomization portion of the parent study.

If you give us your permission, we would like to collect extra samples of your blood and marrow at several time points during your participation on the parent trial.

#### C. Why are you doing this study?

We are collecting samples to learn more about how your body responds to the treatment on the parent trial. We will collect samples on 60 patients across all treatment arms. Your participation on this study is expected to last up to 3 years.

#### D. What will happen to me if I join the study?

If you say you want to be in the study, we will ask you for the following samples:

- Bone Marrow Aspirate Samples: About 1 teaspoon of bone marrow will be collected at the following timepoints:
  - Just before you are randomized on the parent trial (about 50-80 days after your bone marrow transplant). This is one teaspoon more of bone marrow being collected at the time of a required bone marrow aspirate being performed as part of the primary trial.
  - o Just before you start your 9<sup>th</sup> Cycle of Maintenance (about 1 year after your bone marrow transplant). This is one teaspoon more of bone marrow being collected at

the time of a required bone marrow aspirate being performed as part of the primary trial.

 If your disease comes back, an additional bone marrow aspirate sample will be collected at that time. This is an additional aspirate not required as part of the primary trial.

#### • Blood Samples:

- About 2 teaspoons of blood will be collected just before you start Cycles 1, 2, and
   4 of Maintenance Therapy. This is extra blood being collected at the time of a required blood sample collection being performed as part of the primary trial.
- o If your disease comes back, about 10 teaspoons of blood will be collected at that time. This is an additional collection not required as part of the primary trial.
- We will also use a portion of the bone marrow aspirate sample that you already provided at the time of agreeing to participate on the BMT CTN 1401 study as part of this research sample study.

#### E. Where will my samples be sent?

Your samples will be sent to a laboratory at Beth Israel Deaconess Medical Center.

All research samples will be tied to a number. This number will not be linked to your name or other identifying information.

## **Statement of Consent for Research Samples**

The purpose of providing blood and bone marrow samples, the procedures involved, and the risks and benefits have been explained to me. I have asked all the questions I have at this time and I have been told whom to contact if I have more questions. I have been told that I will be given a signed copy of this consent form to keep.

I understand that I do not have to allow the use of my blood and bone marrow for this research. If I decide to not let collect research samples now or in the future, it will not affect my medical care in any way.

| I voluntarily agree that my blood, bone marrow, and information | can be used for the study entitled |
|---|---|
| "Characterization of the T cell immune response and myeloma | genomic signature as predictors |
| of immunologic and clinical response". I also understand that | my DNA and health information |
| may or may not be used in genome-wide association studies. | |
| Signature | Date |

#### Supplemental Informed Consent Form to Participate in Research

**Study Title:** VCAN Proteolysis: Investigation of a Potential Novel Immune Biomarker in Myeloma

**Parent Study Title:** Phase II Multicenter Trial of Single Autologous Hematopoietic Cell Transplant Followed by Lenalidomide Maintenance for Multiple Myeloma with or without Vaccination with Dendritic Cell /Myeloma Fusions

#### A. What is this Document?

The purpose of this document is to give you more information on the bone marrow sample study your physician is asking for your consent to join. This document will explain further details of what samples are collected, why they are being collected, and where they are being sent. Details about risks, study participation, and your rights are explained in the primary informed consent form that your doctor already presented to you. If you want to participate in this research you will be asked to sign the primary informed consent form as well as this document.

#### B. Why am I here?

You are being asked to participate in this study because you are participating on BMT CTN 1401 and are approaching the randomization portion of the parent study.

If you give us your permission, we would like to send a portion of a clinical bone marrow sample to study investigators at the time of randomization. The sample we are asking for is part of a clinical sample collection procedure you will have already undergone as part of the parent trial. We will not collect any additional samples as part of this study. We are asking for your consent to ship a portion of this clinical bone marrow sample to a different lab and study it for research purposes.

#### C. Why are you doing this study?

We are collecting bone marrow samples to learn more about how your body responds to the treatment on the parent trial. We will collect samples on 20 patients across all treatment arms. Your participation on this study is expected to last 1 month. We may use data collected on the parent trial for this study for up to 3 years after you are randomized on the parent trial.

#### D. What will happen to me if I join the study?

The bone marrow sample we are asking for is part of a procedure you will already undergo as part of the parent trial. We will not collect any additional samples as part of this study. We are

asking for your consent to ship a portion of this bone marrow sample to a different lab and study it for research purposes.

If you say you want to be in the study, we will not collect any additional samples. The clinical pathology lab at /Institution/ will cut a small piece of your bone marrow biopsy that you provided for the BMT CTN 1401 parent trial and ship it to investigators at University of Wisconsin. If the lab is not able to obtain enough sample from the bone marrow biopsy you provided for the parent trial (BMT CTN 1401), you will not be asked to provide additional samples and you will be removed from the study.

#### E. Where will my samples be sent?

Your samples will be sent to a laboratory at University of Wisconsin.

All research samples will be tied to a number. This number will not be linked to your name or other identifying information.

## **Statement of Consent for Research Samples**

The purpose of providing bone marrow biopsy samples, the procedures involved, and the risks and benefits have been explained to me. I have asked all the questions I have at this time and I have been told whom to contact if I have more questions. I have been told that I will be given a signed copy of this consent form to keep.

I understand that I do not have to allow the use of my bone marrow biopsy samples for this research. If I decide to not let collect research samples now or in the future, it will not affect my medical care in any way. It will also not affect my participation in the Parent Trial.

| I voluntarily agree that my bone marrow biopsy samples and information can be used for the study |
|---|
| entitled "VCAN Proteolysis: Investigation of a Potential Novel Immune Biomarker in Myeloma". |
| I also understand that my DNA and health information may or may not be used in genome-wide |
| association studies. |

| Signature | Date |
|-----------|------|